CLINICAL TRIAL: NCT04101149
Title: Genetiska Orsaker Till familjär Hyperkolesterolemi- Mekanism, Prognos Och Individanpassad Behandling
Brief Title: Genetic Causes of Familial Hypercholesterolemia
Status: Active, not recruiting | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 262231
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for investigation of lipids, electrolytes, markers of inflammation and myocardial injury. Blood samples for extraction of DNA for genetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Patients with high clinical suspicion of familial hypercholesterolemia. No intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
Familial hypercholesterolemia (FH) is a common disease. The genetic background to FH is not yet fully understood. In the present prospective cohort study we aim to study the association between different clinical characteristics, gene mutations and prognosis.

DETAILED DESCRIPTION:
In this prospective observational cohort study of patients with high clinical suspicion of familial hypercholesterolemia (FH) we aim to study the association between different clinical characteristics, gene mutations and prognosis.

The included patients will undergo physical examination and extended blood sampling. DNA will be extracted and used for both whole genome sequencing and investigation of both known- , unknown- and suspected mutations associated with FH.

The patients will be followed in for 15 years in the Swedish patients registry and the Swedish cause of death registry.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 years or older.
2. Clinical suspicion of FH
3. Dutch Lipid Clinic Network Score of at least four or a first grade relative with a genetic deviation that may be associated with FH.

Exclusion Criteria:

1) Age below 8 years.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected FH referred to the cardiac clinic at Orebro University hospital and their first grade relatives.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mutations. | 2 years
  The prevalence of known and newly discovered mutations associated with FH in the study population.

SECONDARY OUTCOMES:
Prognosis, composite endpoint. | 10 years
  Time to death (cardiovascular and total), hospitalization due to acute myocardial infarction, unstable angina, heart failure or stroke.
Prognosis, individual endpoint. | 10 years
  Time to the individual endpoints: death (cardiovascular and total), hospitalization due to acute myocardial infarction, unstable angina, heart failure, stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Nordenskjöld, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided